CLINICAL TRIAL: NCT05723120
Title: Development and Validation of the PHYSIOSCORE to Assess the Complexity Level and Physiotherapy Care in Hospitalized Patients
Brief Title: Development and Validation of the PHYSIOSCORE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Sao Paulo (Other)
Responsible Party: Principal Investigator, Alcino Costa Leme, Head Physiotherapist of Surgical ICU, University of Sao Paulo
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Health Services Research
Other Study IDs: PHYSIOSCORE
Record Dates: First submitted 2023-01-18; First posted 2023-02-10 (Actual); Last update posted 2023-02-10 (Actual); Status verified 2023-02

CONDITIONS: Heart Diseases; Lung Diseases
MeSH Terms: conditions — Heart Diseases; Lung Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Neuromuscular Score (Experimental): Patients undergoing spontaneous ventilation, noninvasive mechanical ventilation, or invasive mechanical ventilation were assessed by two physical therapists with a minimum interval of 15 minutes between them. There was no communication between the physical therapists before, during, or after the assessments. Patients were also evaluated by the EuroSCORE16, SAPS 317, and ARISCAT18 scales. They were evaluated three times during hospitalization: at protocol admission, after five and ten days, or at hospital discharge, whichever occurred first. The surgical patients were also evaluated three times: immediately postoperative, at ICU discharge, and seven days later or at hospital discharge, whichever occurred first.
  In addition, patients' characteristics at hospital admission were also analyzed, including demographic characteristics, clinical signs and symptoms, imaging, laboratory findings, and medical history
  Interventions: Other: Assessment Respiratory and Neuromuscular
- Respiratory Score (Experimental): Patients undergoing spontaneous ventilation, noninvasive mechanical ventilation, or invasive mechanical ventilation were assessed by two physical therapists with a minimum interval of 15 minutes between them. There was no communication between the physical therapists before, during, or after the assessments. Patients were also evaluated by the EuroSCORE16, SAPS 317, and ARISCAT18 scales. They were evaluated three times during hospitalization: at protocol admission, after five and ten days, or at hospital discharge, whichever occurred first. The surgical patients were also evaluated three times: immediately postoperative, at ICU discharge, and seven days later or at hospital discharge, whichever occurred first.
  In addition, patients' characteristics at hospital admission were also analyzed, including demographic characteristics, clinical signs and symptoms, imaging, laboratory findings, and medical history
  Interventions: Other: Assessment Respiratory and Neuromuscular

INTERVENTIONS:
Other: Assessment Respiratory and Neuromuscular — Comparative Score

SUMMARY:
Abstract Background: Several medical scores have been developed to support clinical support and predict complications in hospitalized patients. However, there is no scale for physical therapy (PT) support.

Objetivo: To develop a scale to determine the level of complexity and PT support in hospitalized patients.

Methods: This cross-sectional study was performed in a tertiary hospital and developed in three distinctive phases: scale (PHYSIOSCORE) development, validation, and testing. The development phase was performed with ten senior PTs using the Delphi methodology. The validation and testing phases were performed by assessing 220 patients (n=110 in each phase). The reproducibility was evaluated by re-assessing 110 patients every five days until hospital discharge.

DETAILED DESCRIPTION:
Phase 1. Questionnaire validation construct. The committee comprised ten specialist physical therapists with more than ten years of experience in hospital care. The questionnaires were developed based on variables used in clinical practice. The committee agreed that the scale needed to meet four objectives7: (i) be composed of variables used by physical therapists working in the hospital; (ii) have valid content for hospitalized adult patients8; (iii) be viable9 (fast and easy to use); and (iv) have inter-examiner reliability.

In the first meeting, every committee member was asked to report relevant variables. After that, the committee was asked to classify each informed variable10-13 as unimportant, important, or essential for the physical therapy assessment to provide quality care to the patient during hospitalization. The validity of this construct was performed using the Delphi technique14,15, and the consensus was defined with a minimum percentage of at least 75% agreement as important or essential. Only the items that reached consensus were retained for the second round.

In the second round, the committee members were asked to re-evaluate each item and classify them on a 10-point numerical scale. Where the score 0 represented the item within the normal range and 5, 7, or 10 points, depending on the item analyzed, the condition that most deviated from normality and consequently would result in greater attention and greater complexity of physical therapy care (Appendix B). The consensus was defined with a minimum percentage of at least 75% agreement among the participants for each item.

The final version of the PHYSIOSCORE was composed of 106 items, divided into three domains: respiratory, imaging, and neuromuscular. For patients with spontaneous breathing or noninvasive mechanical ventilation, the PHYSIOSCORE consisted of six items: pulmonary function, pulmonary sound, need for airway clearance, peripheral oxygen saturation (SpO2), respiratory rate (f), and imaging examination. For patients on invasive mechanical ventilation, the PHYSIOSCORE was also composed of six items: pulmonary sound, PaO2/FiO2 ratio, patient-mechanical ventilator interaction, measurements of pulmonary mechanics, need for airway clearance, and imaging examination (Appendix C). The imaging examination was divided into four segments: pulmonary parenchyma, pleura, vascular plot, and expandability (Appendix D).

The neuromuscular evaluation consisted of six items: neuropsychological, muscle strength and tone, postural control, neuromotor coordination, and walking. (Appendix E).

In the third round, the committee reviewed the PHYSIOSCORE, seeking redundancies and ensuring the final writing of all items and domains.

Phase 2. Concordance and Interrater Reliability This phase was performed by another ten physical therapists (not involved in phase 1) with at least five years of experience in the hospital setting. In addition, the online calculator was developed to include the 106 items divided into three main domains of PHYSIOESCORE (http://www.fisioescore.com, in Portuguese). All physical therapists received prior training to standardize the use of the scale.

The interrater agreement and reliability were established following a prospective and observational single-center study. A cohort of 110 patients hospitalized for clinical or surgical cardiac conditions was recruited from March to June 2019. Patients were selected with the following inclusion criteria: age between 18 and 80 years, both sexes, and pre- or postoperative cardiac surgery. The exclusion criteria were as follows: participating in another study, being unable to understand and perform any of the proposed tests, and cardiovascular instability. Before participating in the study, all patients signed a written informed consent form.

Patients undergoing spontaneous ventilation, noninvasive mechanical ventilation, or invasive mechanical ventilation were assessed by two physical therapists with a minimum interval of 15 minutes between them. There was no communication between the physical therapists before, during, or after the assessments. Patients were also evaluated by the EuroSCORE16, SAPS 317, and ARISCAT18 scales. They were evaluated three times during hospitalization: at protocol admission, after five and ten days, or at hospital discharge, whichever occurred first. The surgical patients were also evaluated three times: immediately postoperative, at ICU discharge, and seven days later or at hospital discharge, whichever occurred first.

In addition, patients' characteristics at hospital admission were also analyzed, including demographic characteristics, clinical signs and symptoms, imaging, laboratory findings, and medical history.

Phase 3 Clinical Validation of the Instrument A total of 110 consecutive clinical and surgical patients were selected. Patients inclusion and exclusion criteria were similar to those evaluated in phase 2. This phase was performed in two stages. Initially, the PHYSIOSCORE was applied to assess the level of attention and complexity of physical therapy care by one professional. Then, a second physical therapist with at least five years of experience performed respiratory and neuromuscular physical therapy. The time spent evaluating respiratory and neuromuscular physical therapist care and registering electronic medical records were all timed.

ELIGIBILITY:
Inclusion Criteria

* age between 18 and 80 years
* both sexes
* pre- or postoperative cardiac surgery.

Exclusion Criteria

* participating in another study
* unable to understand and perform any of the proposed tests
* cardiovascular instability.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 220 (Actual)
Dates: Start 2018-01-10 (Actual); Primary Completion 2021-01-10 (Actual); Study Completion 2022-10-10 (Actual)

PRIMARY OUTCOMES:
Respiratory variables | 3 years
  "lung function", "breath sounds", "PaO2/FiO2", and "Chest X-ray"
neuromuscular variables | 3 years
  "muscle strength", "muscle tone" and "postural control"

CONTACTS AND LOCATIONS:
Overall Officials: Alcino C Leme, PhD, Principal Investigator — University of Sao Paulo
Locations (1):
- Alcino Costa Leme, São Paulo, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] 1. Griffith JR, White KR. The revolution in hospital management. J Healthc Manag. 2005;50(3):170-189; discussion 189-190. 2. Ghasemi M, Ghadiri Nejad M, Bagzibagli K. Knowledge Management Orientation: An Innovative Perspective to Hospital Management. Iran J Public Health. 2017;46(12):1639-1645. 3. Masic I, Miokovic M, Muhamedagic B. Evidence based medicine - new approaches and challenges. Acta Inform Med. 2008;16(4):219-225. 4. Tipping CJ, Young PJ, Romero L, Saxena MK, Dulhunty J, Hodgson CL. A systematic review of measurements of physical function in critically ill adults. Critical care and resuscitation : journal of the Australasian Academy of Critical Care Medicine. 2012;14(4):302-311. 5. Fernandes LEMea. Recursos humanos em hospitais estaduais gerenciados por organizações sociais de saúde: a lógica do privado. Educação e Saúde. 2018;v. 16(n. 3):955-973. 6. Katia de Miranda Avena RPA. CONTRIBUTION OF MANAGEMENT EDUCATION: CHALLENGES OF THE PHYSIOTHERAPIST TO COMPLY WITH THE JOB MARKET DEMANDS. Braz. J. of Develop. 2020;6(8):55974-55987. 7. Mokkink LB, Terwee CB, Knol DL, et al. Protocol of the COSMIN study: COnsensus-based Standards for the selection of health Measurement INstruments. BMC Med Res Methodol. 2006;6:2. 8. Mokkink LB, Terwee CB, Knol DL, et al. The COSMIN checklist for evaluating the methodological quality of studies on measurement properties: a clarification of its content. BMC Med Res Methodol. 2010;10:22. 9. Burns KE, Duffett M, Kho ME, et al. A guide for the design and conduct of self-administered surveys of clinicians. CMAJ : Canadian Medical Association journal = journal de l'Association medicale canadienne. 2008;179(3):245-252. 10. Bickley LS. Bates - Propedêutica Médica. 12ª edição ed: Guanabara Koogan; 2018. 11. Pereira CAC. Medicina Respiratória. Vol 1 e 2. Primeira Edição ed: Atheneu; 2014. 12. Campbell WW. DeJong's O Exame Neurológico. Vol Seventh Edition: Guanabara Koogan; 2014. 13. Kumaran JCaM. Manual de Raios X de Tórax. Vol 4 Edição: Elsevier Editora Ltda; 2017. 14. Diamond IR, Grant RC, Feldman BM, et al. Defining consensus: a systematic review recommends methodologic criteria for reporting of Delphi studies. Journal of clinical epidemiology. 2014;67(4):401-409. 15. Dalkey N, Helmer O. An Experimental Application of the Delphi Method to the Use of Experts. Manage Sci. 1963;9(3):458-467. 16. Nashef SA, Roques F, Sharples LD, et al. EuroSCORE II. European journal of cardio-thoracic surgery : official journal of the European Association for Cardio-thoracic Surgery. 2012;41(4):734-744; discussion 744-735. 17. Moreno RP, Metnitz PG, Almeida E, et al. SAPS 3--From evaluation of the patient to evaluation of the intensive care unit. Part 2: Development of a prognostic model for hospital mortality at ICU admission. Intensive care medicine. 2005;31(10):1345-1355. 18. Bisbe E, Sabate S, Castillo J, Basora M, Canet J. Postoperative complications related to allogeneic transfusion in major surgery. The multicenter, prospective study ARISCAT. European journal of anaesthesiology. 2010;27(1):110-110. 19. Zegers M, de Bruijne MC, Wagner C, Groenewegen PP, van der Wal G, de Vet HC. The inter-rater agreement of retrospective assessments of adverse events does not improve with two reviewers per patient record. Journal of clinical epidemiology. 2010;63(1):94-102. 20. Warrens MJ. Chance-corrected measures for 2 x 2 tables that coincide with weighted kappa. Br J Math Stat Psychol. 2011;64(Pt 2):355-365. 21. Malmoon Z, Tourani S, Maleki M, Jafari M. Future competencies for hospital management in developing countries: Systematic review. Med J Islam Repub Iran. 2020;34:15. 22. Franco SS, Malbouisson LMS, Grinberg M, Feltrim MIZ. A propose of pulmonary dysfunction stratification after valve surgery by physiotherapeutic assistance level. Rev Bras Cir Cardiov. 2015;30(2):188-197. 23. Schweickert WD, Pohlman MC, Pohlman AS, et al. Early physical and occupational therapy in mechanically ventilated, critically ill patients: a randomised controlled trial. Lancet. 2009;373(9678):1874-1882. 24. Corner EJ, Wood H, Englebretsen C, et al. The Chelsea critical care physical assessment tool (CPAx): validation of an innovative new tool to measure physical morbidity in the general adult critical care population; an observational proof-of-concept pilot study. Physiotherapy. 2013;99(1):33-41. 25. Perme C, Nawa RK, Winkelman C, Masud F. A tool to assess mobility status in critically ill patients: the Perme Intensive Care Unit Mobility Score. Methodist DeBakey cardiovascular journal. 2014;10(1):41-49. 26. Canet J, Mazo V. Postoperative pulmonary complications. Minerva anestesiologica. 2010;76(2):138-143. 27. Canet J, Gallart L, Gomar C, et al. Prediction of postoperative pulmonary complications in a population-based surgical cohort. Anesthesiology. 2010;113(6):1338-1350.